CLINICAL TRIAL: NCT05943041
Title: Open-label, Single-center, Dose-escalation Phase 1 Clinical Study to Evaluate the Safety and Tolerability of GB104, and Explore Gut Microbial Composition in Patients Who Completed Curative Colectomy and Planned Therapy of Colorectal Cancer
Brief Title: Live Biotherapeutic Product GB104 Phase 1 Study in Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GILongevity (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GB-X01-101
Record Dates: First submitted 2023-06-22; First posted 2023-07-12 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Solid Tumor; Colorectal Cancer; Sigmoid Colon Cancer; Rectosigmoid Junction Cancer; Cancer; Rectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Sigmoid Neoplasms; Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Sequential Group Assignment (3+3 model)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- GB104: Dose level 1 (Experimental): Dose escalation cohort includes patients with CRC who completed curative colectomy and planned therapy. 3 to 6 patients will be enrolled per escalating dose levels.
  Interventions: Drug: GB104(Level 1)
- GB104: Dose level 2 (Experimental): Dose escalation cohort includes patients with CRC who completed curative colectomy and planned therapy. 3 to 6 patients will be enrolled per escalating dose levels.
  Interventions: Drug: GB104(Level 2)
- GB104: Dose level 3 (Experimental): Dose escalation cohort includes patients with CRC who completed curative colectomy and planned therapy. 3 to 6 patients will be enrolled per escalating dose levels.
  Interventions: Drug: GB104(Level 3)

INTERVENTIONS:
Drug: GB104(Level 1) — One capsule QD oral administration for 28 days
  Arms: GB104: Dose level 1
Drug: GB104(Level 2) — Three capsules QD oral administration for 28 days
  Arms: GB104: Dose level 2
Drug: GB104(Level 3) — Five capsules QD oral administration for 28 days
  Arms: GB104: Dose level 3

SUMMARY:
Prospective, open label, multi-dose, sequential dose escalation, single-center, Phase 1 trial

DETAILED DESCRIPTION:
This is a single center, open-label, phase 1 study to evaluate the safety and tolerability of GB104 and explore gut microbial composition in patients with colorectal cancer who completed standard treatment including curative colectomy with or without full-cycle adjuvant chemotherapy. GB104 is a live biotherapeutic product consisting of a lyophilized formulation of a single strain of bacterium. The dosing regimen for the study involves the oral administration of the experimental drug once a day.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who sign on an informed consent form willingly
2. Subjects who have histological and radiological diagnosis of colorectal cancer
3. Males and females aged between 19 and 80 years at the time of screening
4. Subjects who have undergone radical colectomy and received the following treatments before participating in the clinical trial, and have completed the specified period:

   * Subjects who have received adjuvant chemotherapy, radiotherapy, or concurrent chemoradiotherapy and have completed 3 months since the last treatments
   * Subjects who have not received any adjuvant therapy and have completed 3 months from the radical colectomy
   * Subjects who have undergone stoma closure and have completed 3 months after stoma closure
5. Subjects who have received standard treatment for colorectal cancer without disease progression or recurrence until the first administration of GB104
6. Subjects who have received adjuvant chemotherapy or radiation therapy, and have completed 3 months after completing the treatment, and toxicity from previous adjuvant treatment must have recovered to NCI-CTCAE v5.0 grade 1
7. Subjects who have been confirmed to have adequate hematological, renal, and hepatic function at the screening point (laboratory tests may be retested during the screening period)
8. Female subjects of childbearing potential and sexually active men who agree to abstain from sexual activity or use an adequate method of contraception

Exclusion Criteria:

1. Significant cardiac dysfunction, New York Heart Association classification for chronic heart failure III-IV, symptomatic coronary artery disease, significant deep vein thrombosis; myocardial infarction within 6 months
2. Severe active infections that require systemic antibiotics, antifungal agents, antiviral agents, or other medications that cannot be controlled
3. Previous history of immunosuppressant within the 1 month of initial administration
4. Known HIV infection, or active infection with hepatitis B or C
5. Subjects who have completed a course of antibiotics within the one month prior to screening

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2023-04-28 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Incidence of DLT(Dose-Limiting Toxicity) at week 4 | 4 weeks
Incidence of Adverse Events from baseline to 8 weeks | assessed up to 8 weeks

OTHER OUTCOMES:
Quantity and persistence of GB104 in fecal sample from baseline to 8 weeks | assessed up to 8 weeks
  analyzed by quantitative PCR
Changes in composition of gut microbiota in fecal samples from baseline to 8 weeks | assessed up to 8 weeks
  analyzed by 16S rRNA gene amplicon sequencing
Changes in immune status from baseline to 8 weeks | assessed up to 8 weeks
  * Immune response activation factors(cytokine)
  * Immunophenotyping of peripheral blood mononuclear cells will be performed by flow cytometry
Changes in quality of life improvement from baseline to 8 weeks | assessed up to 8 weeks
  analyzed by EQ-5D-5L(EuroQoL 5-Dimensions 5-Level) questionnaire
Changes of LARS(Low Anterior Resection Syndrome) score from baseline to 8 weeks | assessed up to 8 weeks
  analyzed by LARS questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Woo Yong Lee, M.D., Ph.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, Gangnam-gu, South Korea

IPD SHARING:
Plan to Share IPD: No